CLINICAL TRIAL: NCT06331728
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study With Single Blind Sentinel Period to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IGNX001 in Peanut-Allergic Participants
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of IGNX001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IgGenix Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IGNX-T1
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, single ascending dose study with single blind sentinel period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: With the exception of the single sentinel participants for each cohort who will be single blinded (participant blinded), the study will be designed as a double-blind study thus the Investigator, site staff (other than pharmacists), sponsor, sponsors delegates (if applicable) and participants are all blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IGNX001 (Experimental): Participants will receive IGNX001 given as a single subcutaneous dose on Day 1.
  Interventions: Drug: IGNX001
- Placebo (Placebo Comparator): Participants will receive IGNX001 placebo given as a single subcutaneous dose on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IGNX001 — IGNX001 given as a single subcutaneous dose on Day 1.
  Arms: IGNX001
Drug: Placebo — Placebo to IGNX001 given as a single subcutaneous dose on Day 1.
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled, single ascending dose clinical trial is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of IGNX001 in peanut-allergic adults and older Adolescents.

ELIGIBILITY:
Key Inclusion Criteria:

* History of physician-diagnosed peanut allergy with clinical reaction to peanut within 2 hours of exposure to peanut or peanut-containing food (within the last 15 years).
* Peanut specific IgE level ≥ 1 kUA/L.
* Positive peanut SPT with wheal diameter ≥ 5 mm.

Key Exclusion Criteria:

* History of severe or life-threatening anaphylaxis requiring intubation or admission to intensive care unit within 1 year prior to Screening.
* Current, or within the past year, treatment with food allergen immunotherapy or participation in a food allergy immunotherapy study.
* Current treatment with aeroallergen immunotherapy, except if on stable monthly maintenance SC aeroallergen immunotherapy.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events | From time of dose until Exit Visit/Early Termination Visit or until AE is resolved or no further follow-up is required, whichever is longer (up to 13 weeks).
  Treatment emergent adverse events (TEAE) are undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. All adverse events will be captured and assessed.
Incidence of Serious Adverse Events and Suspected Unexpected Serious Adverse Reactions | From consent until Exit Visit/Early Termination Visit or until SAE is resolved or no further follow-up is required, whichever is longer (up to 13 weeks).
  A serious adverse events is an adverse event that meets the criteria of being serious as determined by the Investigator. Suspected unexpected serious adverse reactions is an event assessed as serious, related to study product, and unexpected, which are subject to expedited reporting to regulatory authorities and study Investigators.
Number of Participants with Clinically significant Changes from Baseline - Hematology | Assessed at Screening, Days 1, 2, 4, 8, 15, 29, 43, 57, 71, and 85 (up to 25 weeks).
  The following list of attributes will be assessed: Hemoglobin, hematocrit, erythrocytes, reticulocytes, platelets, leukocytes (white blood cells), differentials (counts): neutrophils, basophils, eosinophils, lymphocytes, and monocytes
Number of Participants with Clinically Significant Changes from Baseline - Chemistry | Assessed at Screening, Days 1, 2, 4, 8, 15, 29, 43, 57, 71, and 85 (up to 25 weeks).
  The following list of attributes will be assessed: Aspartate aminotransferase, alanine aminotransferase, total and conjugated bilirubin, alkaline phosphatase, gamma-glutamyl-transferase, creatine phosphokinase, albumin, creatinine, blood urea nitrogen, total protein, sodium, chloride, calcium, phosphate, potassium, triglycerides, total cholesterol, glucose.
Number of Participants with Clinically Significant Changes from Baseline - 12-lead ECGs for HR, PR, QRS, QT, RR and QTcF, and information on T- and U-waves | Assessed at Screening, Days 1, 15, and 85 (up to 25 weeks).
  All ECGs will be obtained in supine position following a 10-minute rest. Any clinically significant ECG abnormalities will be captured and reported.
Number of Participants with Clinically Significant Changes from Baseline - Physical Examinations | Assessed at Screening, Days 1, 2, 4, 8, 15, 29, 43, 57, 71, and 85 (up to 25 weeks).
  Complete physical examinations include general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.
  Body weight (kilogram) and height (meter) will be obtained with the participant's shoes and jacket or coat removed. Body mass index is calculated by dividing the participant's body weight in kilograms by the participant's height in meters, squared (kg/m2).

SECONDARY OUTCOMES:
Concentration of IGNX001 in the Plasma | Assessed at Days 1, 2, 4, 8, 15, 29, 43, 57, 71 and 85 (up to 13 weeks).
  Plasma concentrations of IGNX001 will be measured by a specific and validated immunoassay.
Measurement of Area under the Plasma/Serum Concentration Curve (AUC) | Assessed at Days 1, 2, 4, 8, 15, 29, 43, 57, 71 and 85 (up to 13 weeks).
  PK parameters will be computed using non-compartmental analysis (NCA) using the software WinNonlin (Certara, Inc. Princeton, New Jersey). Actual times for drug administration and blood sampling will be used to compute PK parameters.
  * AUClast - Area under the concentration-time curve from time zero to the time point of the last reportable concentration (Cplast).
  * AUCtotal - Area under the concentration-time curve from time zero to infinity, computed as AUCtotal = AUClast + Cplast/lambda where lambda is the slope of the regression curve used to compute half-life.
  * AUC extrapolated - the percent of AUCtotal extrapolated beyond the last reportable concentration (Cplast). AUC extrapolated = 100 x (Cplast/lambda)/AUCtotal.
  * AUCx-y - Partial area under the concentration-time curve from time x to time y. More than 1 partial AUC will be computed as feasible.
Peak Serum Concentration (Cmax) | Assessed at Days 1, 2, 4, 8, 15, 29, 43, 57, 71 and 85 (up to 13 weeks).
  PK parameters will be computed using non-compartmental analysis (NCA) using the software WinNonlin (Certara, Inc. Princeton, New Jersey). Actual times for drug administration and blood sampling will be used to compute PK parameters.
  Cmax - Peak concentration
Time to Peak Serum Concentration (Tmax) | Assessed at Days 1, 2, 4, 8, 15, 29, 43, 57, Day 71 and 85 (up to 13 weeks).
  PK parameters will be computed using non-compartmental analysis (NCA) using the software WinNonlin (Certara, Inc. Princeton, New Jersey). Actual times for drug administration and blood sampling will be used to compute PK parameters.
  Tmax - Time of Cmax
Elimination Half-life (t1/2) | Assessed at Days 1, 2, 4, 8, 15, 29, 43, 57, 71 and 85 (up to 13 weeks).
  PK parameters will be computed using non-compartmental analysis (NCA) using the software WinNonlin (Certara, Inc. Princeton, New Jersey). Actual times for drug administration and blood sampling will be used to compute PK parameters.
  Half-life for each phase of decline in concentrations - Computed from the ln-linear slope (lambda) of the regression on the terminal phase of the concentration-time curve. Half-life = ln(2)/lambda. Rules for acceptance of half-life to be based on robustness of the correlation coefficient for the ln-linear regression to be defined in the SAP.
Changes Over Time to Anti-drug Antibodies | Assessed at Day 1, Day 15, Day 29, Day 57 and 85 (up to 13 weeks).
  The detection and characterization of antibodies to IGNX001 will be performed using a validated assay method under the supervision of the Sponsor.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - St Vincent's Sydney, Darlinghurst, New South Wales
  - Monash Health, Sleep, Allergy, and Immunology, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia